CLINICAL TRIAL: NCT03319901
Title: A Phase Ib Study of the Combination of Venetoclax With Chemotherapy as Frontline Therapy in Older Patients and Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia
Brief Title: Venetoclax and Chemotherapy as Frontline Therapy in Older Patients and Patients With Relapsed/Refractory ALL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Marlise Luskin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-648
Record Dates: First submitted 2017-09-28; First posted 2017-10-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Leukemia
Keywords: Leukemia
MeSH Terms: conditions — Leukemia | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax + Chemotherapy (Experimental): * Venetoclax is administered orally once daily for 21 days in each cycle
  * Standard Chemotherapy will be administered every 28 days
  Interventions: Drug: Venetoclax; Drug: Standard Chemotherapy

INTERVENTIONS:
Drug: Venetoclax — Venetoclax is an inhibitor of Bcl-2. Bcl-2 is critical for keeping cancer cells alive.
  By inhibiting Bcl-2, venetoclax promotes cancer cell death.
  Other Names: ABT199
Drug: Standard Chemotherapy — Standard treatment of chemotherapy is administered

SUMMARY:
This research study is studying a medication called Venetoclax and a chemotherapy regimen as a possible treatment for Acute Lymphoblastic Leukemia.

The drugs involved in this study are:

* Venetoclax
* Standard Chemotherapy (which includes cyclophosphamide, vincristine, doxorubicin, dexamethasone, methotrexate, 6-mercaptopurine, etoposide, and cytarabine

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and drug combination and also tries to define the appropriate dose of the investigational drug and drug combination to use for further studies. "Investigational" means that the drug and drug combination is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved Venetoclax for this specific disease, but it has been approved for other uses.

Venetoclax is an inhibitor of Bcl-2. Bcl-2 is critical for keeping cancer cells alive.

By inhibiting Bcl-2, venetoclax promotes cancer cell death. This drug is currently being used in other clinical trials for people with certain types of leukemia, lymphoma, and multiple myeloma. There is some evidence from those and other laboratory trials that venetoclax may kill cancer cells and cause tumors to shrink.

In this research study, the investigators are investigating how safe the combination of Venetoclax and standard chemotherapy is and how it affects this disease.. The participant will be given Venetoclax alone first and the standard chemotherapies will be given in combination. This study aims to provide information to help determine the dose of Venetoclax , in combination with standard chemotherapy, affects this disease the best and which dose is the safest.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated acute lymphoblastic leukemia (B-cell or T-cell)
* Bone marrow involvement with ≥20% lymphoblasts
* Age ≥ 60 Years

OR

* Patients with relapsed or refractory acute lymphoblastic leukemia (B-cell or T-cell) defined as receiving one or more cytotoxic containing regimens
* Bone marrow involvement with ≥5% lymphoblasts
* Age ≥ 18 Years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Refer to Appendix D)
* Adequate organ function

  * Serum total bilirubin ≤1.5 x upper limit of normal (ULN) or ≤3 x ULN for patients with Gilbert's disease
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 x ULN, unless clearly due to disease involvement
  * Creatinine clearance >50 mL/min (calculated according to institutional standards or using Cockcroft-Gault or Modification of Diet in Renal Disease (MDRD) formula)
* Women of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (β-hCG) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use an effective contraception method during the study and for 30 days following the last dose of study drug. Women of non- childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy. Men who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days following the last dose of study drug
* Patients or their legally authorized representative must provide written informed consent

Exclusion Criteria:

* Ph-positive ALL, Burkitt's leukemia/lymphoma, or lymphoblastic lymphoma
* Patient is pregnant or breastfeeding
* Patients with uncontrolled infection
* Hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
* Major surgery or radiation therapy within 4 weeks prior to the first study dose
* Systemic chemotherapy/radiotherapy/investigational therapy within 14 days (with the exception of hydroxyurea and/or dexamethasone, or one dose of cytarabine) prior to starting therapy
* Symptomatic or untreated leptomeningeal disease or spinal cord compression
* Patients with active heart disease (New York Heart Association (NYHA) class 3-4 as assessed by history and physical examination, unstable angina/stroke/myocardial infarction within the last 6 months)
* Patients with a cardiac ejection fraction (as measured by either Multi Gated Acquisition (MUGA) or echocardiogram (EKG)) <40%
* History of another primary invasive malignancy that has not been definitively treated or in remission for at least 2 years. Patients with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses)
* Concurrent use of warfarin
* Received Cytochrome P450 3A (CYP3A) inhibitors (such as fluconazole, ketoconazole, voriconazole, and clarithromycin) within 3 days of starting venetoclax; received strong CYP3A inducers (such as rifampin, rifabutin, phenytoin, carbamazepine, and St. John's Wort) within 3 days of starting venetoclax
* Consumed grapefruit, grapefruit products, Seville oranges, or star fruit within 3 days prior to starting venetoclax
* Prior treatment with venetoclax
* Malabsorption syndrome or other conditions that preclude enteral route of administration
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 2 years
  To determine the maximum tolerated dose (MTD) of venetoclax in combination with chemotherapy in patients with newly diagnosed Acute Lymphoblastic Leukemia (ALL)

SECONDARY OUTCOMES:
To Evaluate The Safety of the Combination | 2 years
  To evaluate the safety of this combination in a dose expansion cohort.
  The proportion of patients having a grade 3 or higher adverse event will be estimated with a 95% confidence interval in the expansion cohort.
Complete Response | 2 years
  To determine the efficacy: complete response (CR) with incomplete marrow recovery (CRi) of venetoclax in combination with chemotherapy in patients with newly diagnosed ALL
Progression Free Survival | 2 years
  To determine the duration of response: progressive-free survival (PFS) and overall survival (OS) of venetoclax in combination with chemotherapy in patients with newly diagnosed ALL
Overall Survival | 2 years
  To determine the duration of response: progressive-free survival (PFS) and overall survival (OS) of venetoclax in combination with chemotherapy in patients with newly diagnosed ALL
Minimal Residual Disease | 2 years
  To determine the rate of minimal residual disease (MRD) negativity in patients achieving CR/CRi and its correlation with disease-free survival (DFS) and OS
Disease Free Survival | 2 years
  To determine the rate of minimal residual disease (MRD) negativity in patients achieving CR/CRi and its correlation with disease-free survival (DFS) and OS
Change in expression of BCL-2 family proteins: BCL-2 | 2 years
  To measure expression and function of Bcl-2 family proteins and its modulation by venetoclax in ALL blasts.
  The change in expression of BCL-2 family proteins from baseline to the time of each response assessment will be measured including BCL-2 and summary statistics including the median and interquartile range of the change will be reported for all patients in the expansion cohort and also summarized for those achieving a CR/CRi and those patients who do not achieve a CR/CRi.
  This is based on section 9.1: We plan to collect bone marrow and peripheral blood samples at baseline, at the time of clinical response assessment and at the time of progression for correlative studies. These will be done in the laboratory of Dr. Marina Konopleva at MDACC and Dr. Tony Letai at DFCI.
Change in expression of BCL-2 family proteins: BCL-XL | 2 years
  To measure expression and function of Bcl-2 family proteins and its modulation by venetoclax in ALL blasts.
  The change in expression of BCL-2 family proteins from baseline to the time of each response assessment will be measured including BCL-XL and summary statistics including the median and interquartile range of the change will be reported for all patients in the expansion cohort and also summarized for those achieving a CR/CRi and those patients who do not achieve a CR/CRi.
  This is based on section 9.1: We plan to collect bone marrow and peripheral blood samples at baseline, at the time of clinical response assessment and at the time of progression for correlative studies. These will be done in the laboratory of Dr. Marina Konopleva at MDACC and Dr. Tony Letai at DFCI.
Change in expression of BCL-2 family proteins: MCL-1 (anti-apoptotic) | 2 years
  To measure expression and function of Bcl-2 family proteins and its modulation by venetoclax in ALL blasts.
  The change in expression of BCL-2 family proteins from baseline to the time of each response assessment will be measured including MCL-1 (anti-apoptotic) and summary statistics including the median and interquartile range of the change will be reported for all patients in the expansion cohort and also summarized for those achieving a CR/CRi and those patients who do not achieve a CR/CRi.
  This is based on section 9.1: We plan to collect bone marrow and peripheral blood samples at baseline, at the time of clinical response assessment and at the time of progression for correlative studies. These will be done in the laboratory of Dr. Marina Konopleva at MDACC and Dr. Tony Letai at DFCI.
Change in expression of BCL-2 family proteins: BCL-2 homology 3 (BH3) | 2 years
  To measure expression and function of Bcl-2 family proteins and its modulation by venetoclax in ALL blasts.
  The change in expression of BCL-2 family proteins from baseline to the time of each response assessment will be measured including BCL-2 homology 3 (BH3) and summary statistics including the median and interquartile range of the change will be reported for all patients in the expansion cohort and also summarized for those achieving a CR/CRi and those patients who do not achieve a CR/CRi.
  This is based on section 9.1: We plan to collect bone marrow and peripheral blood samples at baseline, at the time of clinical response assessment and at the time of progression for correlative studies. These will be done in the laboratory of Dr. Marina Konopleva at MDACC and Dr. Tony Letai at DFCI.
Change in expression of BCL-2 family proteins: BIM | 2 years
  To measure expression and function of Bcl-2 family proteins and its modulation by venetoclax in ALL blasts.
  The change in expression of BCL-2 family proteins from baseline to the time of each response assessment will be measured including BIM and summary statistics including the median and interquartile range of the change will be reported for all patients in the expansion cohort and also summarized for those achieving a CR/CRi and those patients who do not achieve a CR/CRi.
  This is based on section 9.1: We plan to collect bone marrow and peripheral blood samples at baseline, at the time of clinical response assessment and at the time of progression for correlative studies. These will be done in the laboratory of Dr. Marina Konopleva at MDACC and Dr. Tony Letai at DFCI.
Change in expression of BCL-2 family proteins: BID | 2 years
  To measure expression and function of Bcl-2 family proteins and its modulation by venetoclax in ALL blasts.
  The change in expression of BCL-2 family proteins from baseline to the time of each response assessment will be measured including BID and summary statistics including the median and interquartile range of the change will be reported for all patients in the expansion cohort and also summarized for those achieving a CR/CRi and those patients who do not achieve a CR/CRi.
  This is based on section 9.1: We plan to collect bone marrow and peripheral blood samples at baseline, at the time of clinical response assessment and at the time of progression for correlative studies. These will be done in the laboratory of Dr. Marina Konopleva at MDACC and Dr. Tony Letai at DFCI.
Change in expression of BCL-2 family proteins: BAD | 2 years
  To measure expression and function of Bcl-2 family proteins and its modulation by venetoclax in ALL blasts.
  The change in expression of BCL-2 family proteins from baseline to the time of each response assessment will be measured including BAD and summary statistics including the median and interquartile range of the change will be reported for all patients in the expansion cohort and also summarized for those achieving a CR/CRi and those patients who do not achieve a CR/CRi.
  This is based on section 9.1: We plan to collect bone marrow and peripheral blood samples at baseline, at the time of clinical response assessment and at the time of progression for correlative studies. These will be done in the laboratory of Dr. Marina Konopleva at MDACC and Dr. Tony Letai at DFCI.
Change in expression of BCL-2 family proteins: NOXA | 2 years
  To measure expression and function of Bcl-2 family proteins and its modulation by venetoclax in ALL blasts.
  The change in expression of BCL-2 family proteins from baseline to the time of each response assessment will be measured including NOXA and summary statistics including the median and interquartile range of the change will be reported for all patients in the expansion cohort and also summarized for those achieving a CR/CRi and those patients who do not achieve a CR/CRi.
  This is based on section 9.1: We plan to collect bone marrow and peripheral blood samples at baseline, at the time of clinical response assessment and at the time of progression for correlative studies. These will be done in the laboratory of Dr. Marina Konopleva at MDACC and Dr. Tony Letai at DFCI.
Change in expression of BCL-2 family proteins: PUMA | 2 years
  To measure expression and function of Bcl-2 family proteins and its modulation by venetoclax in ALL blasts.
  The change in expression of BCL-2 family proteins from baseline to the time of each response assessment will be measured including PUMA and summary statistics including the median and interquartile range of the change will be reported for all patients in the expansion cohort and also summarized for those achieving a CR/CRi and those patients who do not achieve a CR/CRi.
  This is based on section 9.1: We plan to collect bone marrow and peripheral blood samples at baseline, at the time of clinical response assessment and at the time of progression for correlative studies. These will be done in the laboratory of Dr. Marina Konopleva at MDACC and Dr. Tony Letai at DFCI.
Change in expression of BCL-2 family proteins: HRK (pro-apoptotic) | 2 years
  To measure expression and function of Bcl-2 family proteins and its modulation by venetoclax in ALL blasts.
  The change in expression of BCL-2 family proteins from baseline to the time of each response assessment will be measured including HRK (pro-apoptotic) and summary statistics including the median and interquartile range of the change will be reported for all patients in the expansion cohort and also summarized for those achieving a CR/CRi and those patients who do not achieve a CR/CRi.
  This is based on section 9.1: We plan to collect bone marrow and peripheral blood samples at baseline, at the time of clinical response assessment and at the time of progression for correlative studies. These will be done in the laboratory of Dr. Marina Konopleva at MDACC and Dr. Tony Letai at DFCI.

CONTACTS AND LOCATIONS:
Overall Officials: Marlise Luskin, MD, MSCE, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
  - Intermountain LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luskin MR, Shimony S, Keating J, Winer ES, Garcia JS, Stone RM, Jabbour E, Flamand Y, Stevenson K, Ryan J, Zeng Z, Letai A, Konopleva M, Jain N, DeAngelo DJ. Venetoclax plus low-intensity chemotherapy for adults with acute lymphoblastic leukemia. Blood Adv. 2025 Feb 11;9(3):617-626. doi: 10.1182/bloodadvances.2024014405. PMID 39546748